CLINICAL TRIAL: NCT00748423
Title: Bicentric Study of the Effect of Inhaled Nitric Oxide Compared to Placebo in Acute Chest Syndrome of Adult Sickle Cell Patients
Brief Title: Effect of Inhaled Nitric Oxide in Acute Chest Syndrome (INOSTA Study)
Acronym: INOSTA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060701
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
Keywords: Inhaled drug; Acute lung injury; Nitric oxide; Sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome; Acute Lung Injury | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nitric Oxide in nitrogen
  Interventions: Drug: Nitric Oxide
- 2 (Placebo Comparator): Nitrogen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — NO in inhalation for 3 days
  Arms: 1
Drug: Placebo — Placebo in inhalation for 3 days
  Other Names: "Nitrogen" placebo
  Arms: 2

SUMMARY:
Acute chest syndrome (ACS) is a frequent and potentially life-threatening pulmonary illness. It is a complication of sickle cell disease and is the leading cause of death from this disease in adults. Several pathologic processes are recognized causes of ACS, including infectious diseases, hypoventilation secondary to chest pain, in situ thrombosis and pulmonary fat embolism. Inhaled nitric oxide (iNO) has been shown to be a pulmonary vasodilatator with minimal systemic effects and has also been shown to improve gas exchange in both animal and human acute lung injury (ALI).

The combined effects of iNO gas of improving pulmonary ventilation to perfusion matching, reducing alveolar and systemic inflammation, modulate the course of acute chest syndrome, which combine the physiopathology of vaso-occlusive crisis and acute lung injury.

We hypothesise inhaled NO will improve oxygenation and clinical outcome of sickle cell disease patients with acute chest syndrome.

DETAILED DESCRIPTION:
Objectives: To compare the outcome and duration of acute chest syndrome (ACS) in patients with sickle cell disease (SCD) treated with iNO to that of similar episodes experienced by patients which receive a placebo.

Study design: Bi-center, prospective, randomized, controlled clinical trial

* Enrollment: 24 months
* Patients will be treated for 72 hours
* Patients will be followed for 15 days or until discharged home

Sample size:

* The study will accrue a maximum of 240 patients
* Progress of the trial will be reviewed by an independent data and safety monitoring committee to determine if randomization should stop for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease (Hemoglobin genotypes characterized by standard procedures as homozygous hemoglobin SS, hemoglobin SC, and S beta thalassemia)
* Diagnosis of acute chest syndrome based on the presence of fever, dyspnea or chest pain, associated with new pulmonary infiltrates on chest X-ray

Exclusion Criteria:

* Patient has been hospitalised < 14 days ago
* Patients presenting with clinically diagnosed bacterial infections
* Patients who have received an exchange transfusion in the last 30 days or are in a transfusion program.
* Current pregnancy or lactation
* Patient who is currently enrolled in any other investigational drug study
* Previous participation in this study
* Any of the following medical conditions:

  * Immediate need of ventilatory support wih orotracheal intubation
  * Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with treatment failure | at day 3

SECONDARY OUTCOMES:
Proportion of hypoxemic patients defined by a PaO2/FiO2 ratio < 300 | at day 3
Variation of pulmonary arterial systolic pressure evaluated by echocardiography | at day 1, day 3 and end of study
Length of hospitalisation | from day 0 to day 15 (max)
Pain assessment and the cumulative dose of parenteral opioids per body weight | during the first three days and during entire hospitalization
Proportion of patients requiring transfusion therapy (simple or exchange) | from day 1 to end of study

CONTACTS AND LOCATIONS:
Overall Officials: MAITRE Bernard, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Réanimation Médicale, Hôpital A Chenevier-H Mondor, Créteil, France

REFERENCES:
- [Derived] Maitre B, Djibre M, Katsahian S, Habibi A, Stankovic Stojanovic K, Khellaf M, Bourgeon I, Lionnet F, Charles-Nelson A, Brochard L, Lemaire F, Galacteros F, Brun-Buisson C, Fartoukh M, Mekontso Dessap A. Inhaled nitric oxide for acute chest syndrome in adult sickle cell patients: a randomized controlled study. Intensive Care Med. 2015 Dec;41(12):2121-9. doi: 10.1007/s00134-015-4060-2. Epub 2015 Oct 2. PMID 26431718